CLINICAL TRIAL: NCT03024593
Title: An Examination of the Effects of Health-related Internet Use in Individuals With Pathological Health Anxiety in a Randomized Controlled Trial
Brief Title: An Examination of the Effects of Health-related Internet Use in Individuals With Pathological Health Anxiety
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Johannes Gutenberg University Mainz (Other)
Collaborators: University of Cologne (Other)
Responsible Party: Principal Investigator, Sandra K. Hamann, Principal Investigator, Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Parallel | Purpose: Basic Science
Other Study IDs: C1-L
Record Dates: First submitted 2017-01-05; First posted 2017-01-19 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Hypochondriasis
Keywords: Cyberchondria; health-related internet use; pathological health anxiety
MeSH Terms: conditions — Hypochondriasis | interventions — Health

ARMS (2):
- Searching condition (Experimental): To simulate participants' natural behavior they are requested to search online for personally relevant health or illness information in their usual manner. By doing so their attentional focus lies on the searching process and the information they obtain.
  Interventions: Behavioral: Health- and illness-related internet use
- Waiting condition (i.e. non- searching, no distraction) (No Intervention): Participants are requested to do nothing and not to distract themselves by reading or using their smartphone for instance. By doing so, it is expected that their attentional focus lies on their induced worries and symptoms.

INTERVENTIONS:
Behavioral: Health- and illness-related internet use
  Arms: Searching condition

SUMMARY:
The purpose of the current study is to examine the effects of health-related internet use on affect, health anxiety and symptom severity in individuals with pathological levels of health anxiety. The present randomized controlled study compares an online medical searching condition with a waiting (i.e. non-searching) condition to manipulate the attentional focus. After an induction of health anxiety using the Autobiographical Emotional Memory Task the participants in the searching condition go online and search for subjectively relevant health information (external focus of attention). Individuals in the waiting (i.e. non-searching) condition are requested to do nothing and not to distract themselves (internal focus of attention).

DETAILED DESCRIPTION:
The internet is a popular method for obtaining information. Increasingly, it is also used to answer medical and health related questions, because compared to other methods (e.g. going to the library or visiting a doctor) it has a number of advantages to offer like low costs, availability, easy accessibility, anonymity, and great diversity of information types and sources. 60 to 80 percent of internet users search online for medical information. In this context the term "cyberchondria" was coined in the media to describe the potentially detrimental effects of this behavior. The first studies in this field using self-report retrospective data showed that individuals with elevated levels of health anxiety seem to make increased use of the internet for this purpose and it seems to maintain health anxiety in the long-term. However, up until today little is known about the consequences of this behavior and the maintaining mechanism.

This randomized controlled experimental study investigates the effects of health-related internet use on affect, symptom severity and health anxiety in individuals with pathological health anxiety. Participants will first undergo a baseline assessment. After that health anxiety is induced using the Autobiographical Emotional Memory Task and participants complete another assessment. Then participants are randomly assigned to either an online medical searching condition (experimental group, EG) or a non-searching condition (control group, CG) to manipulate attentional focus. The EG is requested to search online for health information (external focus of attention), the CG is requested to do nothing and not to distract themselves (internal focus of attention). Then another assessment is completed and the treatment groups are compared regarding the effects on affect, symptom severity and health anxiety. Besides examining these effects a further aim of this study is to identify the underlying mechanism. Two possibilities are supposed: a) An increase of the variables of interest due to health-related information or b) a decrease due to externalization.

ELIGIBILITY:
Inclusion Criteria:

* Pathological health anxiety according to the criteria of Fink et al. (2004)
* Informed consent
* Sufficient German language skills
* Sufficient skills using a computer, a smartphone and the internet

Exclusion Criteria:

* Suicidal tendency
* Clinical diagnosis of alcohol or drug abuse, acute schizophrenia
* Organic brain disorders
* Impairment of intelligence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Primary Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Change of health anxiety before and after 8 minutes of health-related internet searching or waiting | right before and after 8 minutes of health-related internet searching or waiting
  self-created item
Change of positive and negative affect before and after 8 minutes of health-related internet searching or waiting | right before and after 8 minutes of health-related internet searching or waiting
  Positive Affect Negative Affect Schedule - State (PANAS-State)
Change of symptom severity before and after 8 minutes of health-related internet searching or waiting | right before and after 8 minutes of health-related internet searching or waiting
  Checklist for symptoms in daily life (CSD)

SECONDARY OUTCOMES:
Change of health anxiety before and after 10 minutes of anxiety induction | right before and after 10 minutes of anxiety induction
  self-created item
Change of positive and negative affect before and after 10 minutes of anxiety induction | right before and after 10 minutes of anxiety induction
  Positive Affect Negative Affect Schedule - State (PANAS-State)
Change of symptom severity before and after 10 minutes of anxiety induction | right before and after 10 minutes of anxiety induction
  Checklist for symptoms in daily life (CSD)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Witthoeft, Professor, Study Chair — Department of Clinical Psychology, Psychotherapy and Experimental Psychopathology, Johannes Gutenberg University Mainz